CLINICAL TRIAL: NCT06225713
Title: Focused Power Ultrasound Mediated Inferior Perirenal Adipose Tissue Modification Therapy for Non-Alcoholic Fatty Liver Disease: a Randomized Controlled Trial (PARADISE-NAFLD)
Brief Title: Focused Power Ultrasound Mediated Inferior Perirenal Adipose Tissue Modification Therapy for Non-Alcoholic Fatty Liver Disease (PARADISE-NAFLD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Jiangning Hospital of Nanjing Medical University (Other); Suzhou Municipal Hospital (Other)
Responsible Party: Principal Investigator, Xiangqing Kong, Head of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PARADISE-NAFLD
Record Dates: First submitted 2024-01-04; First posted 2024-01-26 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-02

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic Fatty Liver Disease; Focused ultrasound; Novel method
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: This is a randomized, blinded, and sham-control study. The ratio of the intervention group versus sham-control group is 1:1
Who Masked: Participant, Care Provider, Investigator
Masking Description: The masking range includes participants, most researchers (including the study leader; subjects screening researchers; follow-up researchers; sonographers, MR scanners, members of the clinical endpoint identification committee, and etc.) except for the study statistical analysts and the therapy operators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In intervention group, participants will receive the whole peri-renal fat modification therapy (including peri-renal fat ultrasonic measurement and localization, focused ultrasound treatment parameters setting and initiating)
  Interventions: Device: focused power ultrasound mediated inferior perirenal adipose tissue modification
- sham-control group (Sham Comparator): In sham control group, participants will receive the sham control therapy (including peri-renal fat ultrasonic measurement and localization, focused ultrasound treatment parameters setting), however, without initiating the focused ultrasound equipment.
  Interventions: Device: sham-control group

INTERVENTIONS:
Device: focused power ultrasound mediated inferior perirenal adipose tissue modification — This novel focused power ultrasound is an externally delivered, completely noninvasive focused therapeutic ultrasound device. It is capable of focusing the resulting ultrasound beam to a small "cigar"-shaped volume and monitoring the temperature of the target area, which leads to the rapid elevation of the peri-renal adipose tissue temperature and the destruction of target tissue eventually.
  Arms: intervention group
Device: sham-control group — Participants will receive the sham control therapy (including peri-renal fat ultrasonic measurement and localization, focused ultrasound treatment parameters setting), however, without initiating the focused ultrasound equipment.
  Arms: sham-control group

SUMMARY:
This randomized, blinded, sham-control trial aims to evaluate the efficacy and safety of a novel focused power ultrasound mediated inferior perirenal adipose tissue modification therapy for non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Visceral adiposity is closely related to the incidence of non-alcoholic fatty liver disease (NAFLD), and it is also directly associated with liver inflammation and fibrosis. Visceral adiposity, via its unique location and enhanced lipolytic activity, releases toxic free fatty acids, which are delivered in high concentrations directly to the liver and lead to the accumulation and storage of hepatic fat. Furthermore, it has been recognized as an important endocrine organ, and a variety of factors secreted by visceral adiposity may lead to an increased risk of NAFLD.

Peri-renal fat is a special type of visceral adiposity which is different from other type of visceral fat in histology, physiology, and functions. The position of peri-renal fat is more stable than other visceral fat. The investigators found that prophylactic perirenal adipose tissue ablation can prevent the development of NAFLD in mice induced by high fat diets, and also this novel focused power ultrasound can rapidly and efficiently promote the peri-renal adipose tissue fibrosis in the model of swine. Moreover, the investigators performed a single arm, small sample study to investigate the feasibility of the novel focused power ultrasound to modify the inferior peri-renal adipose tissue in NAFLD participants, showing that this kind of method was feasible and safe.

In this study, the investigators aim to further evaluate the efficacy and safety of a novel focused power ultrasound mediated inferior perirenal adipose tissue modification therapy for NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of screening.
* Total liver fat content ≥10% measured by MRI-PDFF.
* Body mass index (BMI) ≥ 25 kg/m^2.
* The anteroposterior, transverse and axial diameters of inferior perirenal fat pad measured by ultrasound should be at least 20mm.
* Participants should be willing to sign the informed consent form of the study.

Exclusion Criteria:

* History of significant alcohol consumption (significant alcohol consumption was defined as more than 140 g/week in females and more than 210 g/week in males in the last 12months before screening, on average).
* Secondary factors causing hepatic steatosis, including viral hepatitis C, autoimmune hepatitis, total parenteral nutrition, celiac disease, Wilson's disease, hypothyroidism, hereditary hemochromatosis, drug factors (amiodarone, glucocorticoids, methotrexate, tamoxifen), etc.
* Complicating other chronic liver diseases, mainly including viral hepatitis, cholestatic liver disease, drug-induced liver injury, etc.
* Weight change >10% in the past 3 months.
* Clinical or pathological diagnosis of cirrhosis.
* NAFLD treatment drugs (such as vitamin E, obecholic acid, thiazolidinediones, etc.) were used within 6 months before enrollment.
* History of bariatric surgery.
* History of kidney and/or surrounding tissue surgery.
* Waist skin infection.
* Urinary stones and/or hematuria (positive for gross hematuria or occult blood).
* Unstable cardiovascular diseases: (1) Myocardial infarction, unstable angina pectoris or cerebrovascular accident occurred in the last 6 months. (2) Persistent atrial fibrillation without anticoagulation. (3) Severe structural heart disease (including valvular heart disease, cardiomyopathy). (4) second degree and above atrioventricular block and/or sick sinus syndrome. (5) Uncontrolled hypertension.
* Type 1 diabetes or uncontrolled hyperglycemia (HBA1c ≥ 9.5%).
* Participants with untreated tumors.
* Laboratory screening results include one or more of the following: (1) Neutrophil absolute value <1.0x10^9/L. (2) Platelet count <100x10^9/L. (3) Hemoglobin <100g/L. (4) Albumin <35g/L. (5) International standard value >1.5. (6) Total bilirubin >1.5 times the upper limit of normal value. (7) The estimated glomerular filtration rate was <60ml/ (minx1.73m^2).
* Participants who are pregnant, breastfeeding or trying to conceive.
* Any contraindication or inability to obtain an MRI.
* Participants who were unable to follow up.
* Any other situation that the investigator considers to be detrimental to the patient's health, hindering the completion of the study, or interfering with the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute Change in Liver Fat Content | From baseline to 3 months post-procedure
  Absolute change in liver fat content assessed by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) at 3-month compared with baseline

SECONDARY OUTCOMES:
Relative Change in Liver Fat Content | From baseline to 3 months post-procedure
  Relative change in liver fat content assessed by MRI-PDFF at 3-month compared with baseline
Proportion of MRI-PDFF Responders | From baseline to 3 months post-procedure
  Proportion of MRI-PDFF responders in two groups at 3-month of treatment. MRI-PDFF responder is defined as a ≥30% relative reduction in MRI-PDFF between baseline and end of treatment
Change in Alanine Aminotransferase (ALT) | From baseline to 3 months post-procedure
  ALT is increased with liver damage. The blood levels of ALT are used to detect liver injury.
Change in Concentration of Cytokeratin-18 | From baseline to 3 months post-procedure
  Change in concentration of cytokeratin-18 in two groups at 3-month of treatment
Change in Liver Stiffness Measurement and Controlled Attenuation Parameter | From baseline to 3 months post-procedure
  Change in liver stiffness measurement and controlled attenuation parameter measured by transient elastography at 3-month of treatment
Change in Enhanced Liver Fibrosis Test | From baseline to 3 months post-procedure
  The markers of fibrosis assessed in this test comprised hyaluronic acid, tissue inhibitor of metalloproteinase 1 and procollagen III N-terminal peptide; these are elevated during fibrogenesis as a result of activation of the hepatic stellate cell.

OTHER OUTCOMES:
Chang in Fasting Lipid Profile | From baseline to 3 months post-procedure
  These include triglycerides, total cholesterol, low-density lipoprotein cholesterol, and high-density lipoprotein cholesterol
Change in Concentration of Fasting Plasma Glucose (FPG) | From baseline to 3 months post-procedure
  Change in concentration of FPG at 3-month compared with baseline
Change in Concentration of Fasting serum insulin (FINS) | From baseline to 3 months post-procedure
  Change in concentration of FINS at 3-month compared with baseline
Change in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) Index | From baseline to 3 months post-procedure
  From the results of FPG and FINS, insulin resistance will be estimated using the HOMA-IR algorithm: HOMA-IR = FPG (mmol/L) × FINS (μU/mL) / 22.5
Change in Percentage of Glycosylated Hemoglobin (Hba1c) | From baseline to 3 months post-procedure
  The structure of Hba1c is relatively stable. Its concentration can effectively reflect the average blood glucose level in the past 8-12 weeks. It should be expressed as a percentage of adult hemoglobin
Change in Body Weight | From baseline to 3 months post-procedure
  Body weight will be measured on a calibrated scale (to the nearest 0.1 kilogram). The measurement will be performed with the study subject in underwear and without shoes; or while wearing minimal indoor clothing
Change in Waist Circumference | From baseline to 3 months post-procedure
  Change in waist circumference at 3-month compared with baseline
Change in Waist to Hip (WTH) Ratio | From baseline to 3 months post-procedure
  The WTH ratio is calculated as the ratio of waist to hip circumference
Change in Office Systolic Blood Pressure | From baseline to 3 months post-procedure
  Change in office systolic blood pressure at 3-month compared with baseline
Change in Office Diastolic Blood Pressure | From baseline to 3 months post-procedure
  Change in office diastolic blood pressure at 3-month compared with baseline
Incidence of Adverse Events (AEs) | From baseline to 3 months post-procedure
  The Incidence AEs will be reported for each arm
Incidence of Severe Adverse Events (SAEs) | From baseline to 3 months post-procedure
  The Incidence SAEs will be reported for each arm

CONTACTS AND LOCATIONS:
Overall Officials: shijing5499@jsph.org.cn Kong, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (3):
- China (3):
  - The Affiliated Jiangning Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - JiangSu Province Hospital / The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu C, Ma Z, Wang Y, Liu X, Tao L, Zheng D, Guo X, Yang X. Visceral adiposity index as a predictor of NAFLD: A prospective study with 4-year follow-up. Liver Int. 2018 Dec;38(12):2294-2300. doi: 10.1111/liv.13941. Epub 2018 Sep 6. PMID 30099825
- [Background] Petta S, Amato MC, Di Marco V, Camma C, Pizzolanti G, Barcellona MR, Cabibi D, Galluzzo A, Sinagra D, Giordano C, Craxi A. Visceral adiposity index is associated with significant fibrosis in patients with non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2012 Jan;35(2):238-47. doi: 10.1111/j.1365-2036.2011.04929.x. Epub 2011 Nov 24. PMID 22117531
- [Background] van der Poorten D, Milner KL, Hui J, Hodge A, Trenell MI, Kench JG, London R, Peduto T, Chisholm DJ, George J. Visceral fat: a key mediator of steatohepatitis in metabolic liver disease. Hepatology. 2008 Aug;48(2):449-57. doi: 10.1002/hep.22350. PMID 18627003